CLINICAL TRIAL: NCT00883142
Title: Functional and Physiological Responses to Lokomat Therapy (Pilot Study)
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B4162C-11
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Spinal Cord Injuries; Multiple Sclerosis; Stroke
Keywords: Lokomat; Suspended walking; Body Weight Supported; Treadmill Training
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and for some muscle biopsy samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Individuals with neurological deficiencies such as those who have spinal cord injury, stroke, traumatic brain injury, Parkinson's disease, and multiple sclerosis often lose their ability to ambulate over ground. Loss of functional mobility not only impedes everyday life, but may also affect many systems and organs in the body. The investigators are interested in obtaining a wide variety of data in order to obtain a better understanding of changes that occur as a result of receiving Lokomat therapy. The investigators will be studying body composition, cardiac, pulmonary, endocrine, metabolic, and molecular changes after a 12-week clinical therapy program.

DETAILED DESCRIPTION:
Description of the Clinical Lokomat Therapy program:

This is a 12-week program with 3 to 5 sessions per week. Each session includes: 15-20 minutes of patient set-up (set-up time becomes about 5 to 10 minutes after a few sessions), 5-10 minutes of warm-up, 20-40 minutes of Lokomat therapy, 5-10 minutes of cool-down, and 5-10 minutes to remove the patient from the system. During the Lokomat sessions, heart rate and blood pressure are monitored by the therapist and recorded. Work performed is measured and recorded in the Lokomat computer for time, speed, amount of weight bearing, and distance.

Description of the Research Component:

A pre and post, prospective study design will be employed. Baseline measurements (Please see below and Table 1 for detailed descriptions) will be performed prior to start of the Lokomat therapy program and then again after completion of the 12-week program. A chart review will be performed at baseline only for documentation of medical history and medications. In a subset of patients a muscle biopsy will be performed for gene expression at baseline and week 12.

As part of Clinical Care, during each of the Lokomat therapy sessions the following information is collected:

1. Work (total time, speed, distance, amount of weight bearing)
2. Heart rate (HR)
3. Blood Pressure (SBP, DBP)
4. Perception of exertion (Borg Scale)
5. Lipid profile (pre and post)
6. Albumin (pre and post)

For Research purposes the following is being proposed:

Review and record work, HR, BP, Borg Scale from all clinical sessions

Baseline and Week 12 measurements (performed on a separate days or prior to the sessions):

1. Resting energy expenditure (REE)
2. Body Composition [dual energy x-ray absorptiometry (DEXA) ) - [scans include total body, dual femur, and the knee], partial body potassium counting (PBKleg), bioelectrical impedance analysis (BIA), anthropometric and skin fold measurements]
3. Fasting blood draw for plasma glucose and insulin (FPG, FPI), lipid profile, testosterone, sex hormone binding globulin (SHBG), insulin-like growth factor 1 (IGF-1), bone markers, coagulation factors, platelet aggregation, 2 hour standard oral glucose tolerance testing (OGTT) with insulin levels.
4. Autonomic and blood pressure regulation studies [resting and tilt table provocation, for heart rate and blood pressure variability (HRV, BPV), arterial blood flow, and venous occlusion]
5. Disability-specific quality of life (QOL) and activities of daily living surveys [GI-Bowel survey, brief pain inventory (BPI), fatigue survey, spasticity scale, mini mental status exam (MMSE)]. These disease-specific QOLs will include the question "How do you rate your general health and well-being over the past week?" A Lickert scale response will be incorporated.
6. Functional Mobility Assessment
7. Muscle biopsy for gene expression (subset of patients only).

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are based on the guidelines set by the clinical Lokomat therapy program.

1. Patients will have been evaluated on the Rehabilitation Service for entry into the clinical therapy program.
2. Any patient who is already eligible for Lokomat therapy is a candidate for this research project.

Exclusion Criteria:

1. Pregnant women
2. History of fractures of the lower extremities
3. Bone density study indicating bone loss greater than 5 standard deviations from normal.
4. Fixed contractures of the ankles, knees or hips
5. Uncontrolled spasticity that significantly interferes with movement of lower extremities.
6. Uncooperative, unmotivated patients or patients whom cannot follow instructions on a consistent basis or communicate effectively with the treating clinicians.
7. Pressure ulcers over the greater trochanters, ischial tuberosities and sacrum.
8. Weight greater than 250 lbs
9. severe orthostatic hypotension (drop in blood pressure more than 30mm Hg when moving from sitting to standing posture)
10. Acute medical illness (i.e. infection)
11. Recently documented DVT in lower extremities
12. SCI ASIA's A and B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lokomat Rehabilitation Clinic
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2006-10; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
This pilot study for power calculations on future studies that will characterize the potential benefits of Lokomat rehabilitation training on cardiovascular function, body composition and endocrine/metabolic function | After completion of 24 clinical Lokomat rehabilitation sessions

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Spungen, EdD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States